CLINICAL TRIAL: NCT06060379
Title: Giochiamo 626 - Gaming for Health and Safety in Workplaces
Acronym: 626 Giochiamo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Mercatorum (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alice Mannocci, Professor, Universitas Mercatorum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6-FIN/RIC2023
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Health; Safety; Workplace
Keywords: Health and Safety workplace

STUDY DESIGN:
Intervention Model Description: The trial consists of three meetings. In the first meeting all enrolled participants will take part in a seminar. Before the seminar starts and at the end, a questionnaire will be administered to them to investigate their prior and acquired knowledge on the subject.
  At the end the participants will be divided into two groups, the control group will not participate in the second phase, the intervention group will be invited to a game meeting. The third meeting will take place days later, where the third and final game will be conducted with the intervention group. At the end of the game, the questionnaire will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention gruop (Experimental): Partecipant will participate in playful encounters
  Interventions: Other: GiochiAMO a 626
- Control group (No Intervention): Subjects will not partecipate in the games

INTERVENTIONS:
Other: GiochiAMO a 626 — The subjects of the intervention group will play three different games: a role-playing game, a card game and a board game.
  Arms: Intervention gruop

SUMMARY:
The aim of the "626 Giochiamo" project is to realise and evaluate the effectiveness of a training course involving the use of games, which helps to convey the basic principles of health and safety in the workplace.

DETAILED DESCRIPTION:
The seminar on health and safety in the workplace and basic principles will be presented to the recruited workers. At the end of the intervention they will be divided into two groups: the control group and the intervention group. The intervention group will be involved in a meeting dedicated to games in three different types, board, card and role-playing games.

A questionnaire on occupational health and safety knowledge will be administered to all study participants before the seminar (T=0), after the seminar (T=1) and after the intervention group has played (T=2).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* No worker

Ages: 17 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of knowledge increased as a result of participation in the games | Participants are assessed by means of a questionnaire administered at the beginning of the trial (t=0), one day after the seminar (t=1) and after one month (t=2).
  Effectiveness is understood as acquiring and increasing knowledge of key concepts on safety in the workplace, the roles of key persons who can influence health and safety, and the tools available for evaluation and monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Mannocci, Principal Investigator — Universitas Mercatorum
Locations (1):
- Alice Mannocci, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
We will share aggregated data, individual data will be submitted upon request by the individual concerned to the Research Contact Person (principal investigator: Alice Mannocci).

REFERENCES:
- [Background] Cocchiara RA, Sestili C, Di Bella O, Backhaus I, Sinopoli A, D'Egidio V, Lia L, Saulle R, Mannocci A, La Torre G. "GiochiAMO," a Gaming Intervention to Prevent Smoking and Alcohol Habits Among Children: A Single-Arm Field Trial. Games Health J. 2020 Apr;9(2):113-120. doi: 10.1089/g4h.2019.0125. Epub 2019 Nov 26. PMID 31770005
- [Background] D'Egidio V, Lia L, Sinopoli A, Backhaus I, Mannocci A, Saulle R, Sestili C, Cocchiara R, Di Bella O, Yordanov T, Mazzacane M, La Torre G. Results of the Italian project 'GiochiAMO' to improve nutrition and PA among children. J Public Health (Oxf). 2021 Jun 7;43(2):405-412. doi: 10.1093/pubmed/fdz129. PMID 31786612
- [Background] La Torre G, Mannocci A, Saulle R, Sinopoli A, D'Egidio V, Sestili C, Manfuso R, Masala D. [GiochiAMO! The protocol of a school based intervention for the promotion of physical activity and nutrition among children]. Clin Ter. 2016 Sep-Oct;167(5):152-155. doi: 10.7417/CT.2016.1947. Italian. PMID 27845482
- [Background] La Torre G, Sinopoli A, Sestili C, D'Egidio V, Di Bella O, Cocchiara RA, Sciarra I, Saulle R, Backhaus I, Mannocci A. "GiochiAMO": a school-based smoking and alcohol prevention program for children - a pilot randomized field trial. Part 2. Ann Ig. 2018 Jul-Aug;30(4):273-284. doi: 10.7416/ai.2018.2219. PMID 29895045
- [Background] La Torre G, Mannocci A, Saulle R, Sinopoli A, D'Egidio V, Sestili C, Manfuso R, Masala D. Improving knowledge and behaviors on diet and physical activity in children: results of a pilot randomized field trial. Ann Ig. 2017 Nov-Dec;29(6):584-594. doi: 10.7416/ai.2017.2187. PMID 29048455
- [Background] La Torre G, D'Egidio V, Sestili C, Cocchiara RA, Cianfanelli S, Di Bella O, Lia L, Dorelli B, Cammalleri V, Backhaus I, Pagano F, Anguissola C, Vitiello A, Carsetti R, Mannocci A, Giochiamo Collaborative Group. ImmunizziAMO: A School-Based Field Trial to Teach New Generations the Importance of Vaccination through Games and to Fight Vaccine Hesitancy in Italy. Vaccines (Basel). 2020 Jun 5;8(2):280. doi: 10.3390/vaccines8020280. PMID 32517111